CLINICAL TRIAL: NCT05412784
Title: Palliative Care Costs for Oncologic and Non-oncologic Patients Under Different Outpatient Management in Catalunya
Brief Title: Palliative Care Costs for Outpatient Setting Management in Catalunya
Acronym: CoCPAC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: 22/006-P
Record Dates: First submitted 2022-05-31; First posted 2022-06-09 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-05

CONDITIONS: Palliative Care; Cost and Cost Analysis; Outpatient
Keywords: Palliative Care [MeSH]; Cost and Cost Analysis [MeSH]; Outpatients [MeSH]

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cost-of-illness studies in palliative care (PC) are a growing area of interest in health economics activity. They are, in part, stakeholders' basis for deciding the allocation of the scarce public and private economic resources. There is no standard methodology to capture the formal and informal costs and expenses that health services and patients and their caregivers make during the PC attention period due to non-standard health services, and data capture approaches.

DETAILED DESCRIPTION:
Methods / Analysis Prospective study on the burden of disease of PC on the outpatient/domiciliary attention. Proposed in three phases: Phase I: Systematic Review of Literature to identify de types of costs and proposed methodologies to identify and determine de economic burden of PC. With collected data, create a questionnaire to register the costs of services covered by the healthcare system and those covered by patients/caregivers (PROSPERO CRD42021250086). Phase II: Questionnaire piloting. Phase III: Transversal study of costs, collecting data from public healthcare billing and patient/caregivers payments to cover PC on selected patients. Final methodologic proposal to study billing/costs of outpatient/domiciliary PC.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of breast, lung, and colorectal neoplasm or Chronic Heart Failure (CHF) or Chronic Obstructive Pulmonary Disease (COPD).
* Patient and caregivers must be able to maintain a 1-hour telephonic interview.
* Patient and caregivers must allow one (1) more telephone call to revise data.

Exclusion Criteria:

* Cases with an open legal process.
* Family/caregivers of patients that can't communicate in fluent Spanish or Catalan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of breast, lung, and colorectal neoplasm or Chronic Heart Failure (CHF) or Chronic Obstructive Pulmonary Disease (COPD), managed in the outpatient/domiciliary scenarios and their families/caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Determination of economic burden (costs) of palliative care in the outpatient context. | 6 months
  Calculation and report the economic burden (i.e., total costs) of outpatient palliative care services, medications and procedures covered and financed by the healthcare system alongside with those covered by the patients and their families/caregivers during the last six (6) months of life (in adult patients with lung, colorectal and breast neoplasms and with terminal cardiac heart failure [CHF] and chronic obstructive pulmonary disease [COPD]).

SECONDARY OUTCOMES:
Type of costs. | 6 months
  Direct, sanitary and non-sanitary costs covered by healthcare system, sanitary and non-sanitary costs covered by patients and families/caregivers and productivity losses due to the patients and families/caregivers to register and measure in a study of costs/economic burden of outpatient palliative care.
Differentiate and compare costs. | 6 months -1 year
  To differentiate and compare direct, sanitary and non-sanitary costs and productivity losses of outpatient palliative care in oncologic and non oncologic patients.

IPD SHARING:
Plan to Share IPD: Undecided
In case the obtained database gives data of public interest, can be used to make parallel analyses, supervised/directed by one of the headline authors.